CLINICAL TRIAL: NCT02781714
Title: Evaluation of an mHealth SMS Dialogue Strategy to Meet Women's and Couples' Postpartum Contraceptive Needs in Kenya
Acronym: Mobile WACh XY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Elizabeth Harrington, Acting Instructor / Family Planning Fellow, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 51125
Record Dates: First submitted 2016-05-14; First posted 2016-05-24 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Contraception; Postpartum Period
Keywords: contraception; postpartum period; mobile health; mHealth; Kenya; couples

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two-way SMS (Experimental): Pre-programmed SMS messages by partner track will be delivered twice weekly to participants in participants' preferred languages from enrollment to 6 months postpartum. They will include a question soliciting a response from the participant(s). Interactive SMS communication will be responded to and managed by the study nurse at each site. Content themes will include: general support/encouragement, postpartum visit reminders, postpartum pregnancy risk and benefits of birth spacing, postpartum contraceptive options and side effects, family planning misconceptions, and couple communication.
  Interventions: Behavioral: Two-way SMS
- Control (No Intervention): The control arm will receive standard education and counseling provided in antenatal care and in postnatal care.

INTERVENTIONS:
Behavioral: Two-way SMS — SMS messages will provide tailored and actionable education, counseling, and reminders specific to antenatal/postpartum timing and partner track. Messages will include questions and prompts; women and their male partners have the option of writing back to a nurse with questions or concerns, who will provide real-time responses via text and/or make referrals to a clinic. Message content will be tailored to women and couples, and will range from health benefits of child spacing and an emphasis on contraceptive options, to the hierarchy of effectiveness and information on specific methods, to simple reminders about postpartum visits.
  Prior to randomization, each enrolled woman will be asked if she has a male partner, and whether she would like to refer her male partner for recruitment and enrollment into the study. The partner tracks are as follows:
  1. Male partner invited to enroll/enrolled
  2. Male partner not invited to enroll
  3. Unpartnered
  Arms: Two-way SMS

SUMMARY:
Meeting women's need for postpartum family planning is has been acknowledged as a global priority in maternal and child health. The prevention of unintended pregnancies in sub-Saharan African countries, which carry the highest global burdens of maternal mortality and HIV infection, is projected to substantially decrease maternal and neonatal morbidity and mortality. Many barriers to contraceptive uptake exist, both within and outside of the postpartum time period, and include socio-cultural, economic, and supply-side factors. Furthermore, while the importance of engaging men in family planning programs has been acknowledged for decades, few interventions have succeeded in increasing male involvement in family planning while maintaining a focus on women's empowerment. Innovative approaches to meeting the family planning needs of women and couples are urgently needed.

Public health interventions are increasingly incorporating mobile health (mHealth) approaches using short message service (SMS) technology in low-income countries, approaches that have demonstrated benefit among various reproductive health outcomes. The investigators hypothesize that personalized, bidirectional SMS dialogue with individual women and couples will increase postpartum contraceptive uptake, thereby decreasing unmet need for family planning in Kenya. The investigators have collaborated with the University of Washington (UW) Department of Computer Science and Engineering (CSE) along with Kenyan telecommunication providers to develop a hybrid messaging system that allows for innovative bidirectional SMS messaging. This system has been used successfully in maternal child health (MCH) clinics in Kenya. In qualitative research, women in Kenya have expressed a strong desire for mHealth support to provide additional education, counseling and reminders to supplement counseling by health workers.

The investigators propose a randomized controlled trial (RCT) comparing the effects of bidirectional SMS dialogue vs. control on highly effective contraceptive use at 6 months postpartum among HIV negative women and couples in Nyanza Province, Kenya. Data from this RCT and accompanying qualitative study will contribute to innovative, scale-able strategies to address unmet need for contraception and increase male involvement in family planning.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant; at least 28 weeks gestation
* HIV negative
* Daily access to a mobile phone
* Planning to stay in area for 6 months postpartum
* Able to read/write or has trusted person to help

Exclusion Criteria:

* Does not meet above criteria

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Highly-effective contraceptive use | 6 months postpartum
  Proportion of participants self-reporting use of oral contraceptive pills, injectable contraception, contraceptive implant, intrauterine device, or male/female sterilization at 6 months postpartum will be compared between arms. Questionnaires will be used to assess this outcome.

SECONDARY OUTCOMES:
Time to contraceptive use | Through study completion (6 months postpartum)
  Time postpartum at which contraceptive use was initiated
Dual contraceptive use | 6 weeks, 14 weeks, and 6 months postpartum
  Percentage of sexual acts in which a condom was used among contraceptive users
Any contraceptive use | 6 weeks, 14 weeks, and 6 months postpartum
  Proportion of participants self-reporting use of any contraceptive method will be compared between arms. This outcome will be assessed with a questionnaire.
Family planning satisfaction questionnaire | 6 weeks, 14 weeks, and 6 months postpartum
  Satisfaction with chosen contraceptive method
Exclusive breastfeeding questionnaire | 6 weeks, 14 weeks, and 6 months postpartum
  Self-reported exclusive breastfeeding

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Ahero sub-County Hospital, Ahero, Kisumu County
  - Bondo County Hospital, Bondo, Siaya County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Harrington EK, Drake AL, Matemo D, Ronen K, Osoti AO, John-Stewart G, Kinuthia J, Unger JA. An mHealth SMS intervention on Postpartum Contraceptive Use Among Women and Couples in Kenya: A Randomized Controlled Trial. Am J Public Health. 2019 Jun;109(6):934-941. doi: 10.2105/AJPH.2019.305051. PMID 31067089